CLINICAL TRIAL: NCT05804604
Title: Serum Concentration of Bone Intake Proteins and Muscle Decay Markers as Risk Factors of Proximal Femur Fractures
Brief Title: Bone Intake Proteins and Muscle Mass Deficiency in Proximal Femur Fractures
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Artur Stolarczyk, Professor, Medical University of Warsaw
Other Study IDs: WarsawMU/FOPF
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-03

CONDITIONS: Femoral Neck Fractures; Pertrochanteric Fracture; Bone Resorption; Bone Loss; Muscle Loss; Muscle Damage
Keywords: proximal femur fracture; femoral neck fracture; pertrochanteric fracture; bone intake proteins; bone resorption; bone loss; muscle damage; muscle loss
MeSH Terms: conditions — Femoral Neck Fractures; Bone Resorption; Bone Diseases, Metabolic; Muscular Atrophy; Proximal Femoral Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Level of bone intake proteins and muscle atrophy marker in patients after proximal femur fracture: Open reduction of femoral neck or pertrochanteric fracture and preoperative analysis of bone intake proteins and muscle atrophy marker serum concentration
  Interventions: Procedure: Surgical treatment of proximal femur fracture and blood sample test
- Level of bone intake proteins and muscle atrophy marker in patients without proximal femur fracture: Control group without a history of proximal femur fracture. Analysis of the bone intake proteins and muscle atrophy marker serum level
  Interventions: Procedure: Blood sample test

INTERVENTIONS:
Procedure: Surgical treatment of proximal femur fracture and blood sample test — Open reduction of femoral neck or pertrochanteric fracture with hemi/total hip arthroplasty or gamma nail. Analysis of serum concentration of: SHBG, CTX - I, CK-MB
  Groups: Level of bone intake proteins and muscle atrophy marker in patients after proximal femur fracture
Procedure: Blood sample test — Analysis of serum concentration of: SHBG, CTX - I, CK-MB
  Groups: Level of bone intake proteins and muscle atrophy marker in patients without proximal femur fracture

SUMMARY:
The aim of this clinical trial is to compare serum concentration of bone intake proteins [ sex hormone-binding globulin (SHBG), cross linked C-telopeptide of type I collagen (CTX-I)] and muscle atrophy marker [creatine kinase (CK-MB)] between patients after the fracture of proximal femur and their age corresponding counterpart without the fracture. The main question it aims to answer is:

• Is the higher concentration of bone intake proteins and muscle atrophy marker a predictive factor of proximal femur fracture?

The part of participants (Group 1) will be hospitalized at the Department of Orthopaedics and Rehabilitation and will undergo a surgical treatment (open reduction of the fracture). The rest (Group 2) will be admitted to the Department of Internal Medicine. Participants of both Groups will have the blood sample test taken, to evaluate and compare the serum concentration of SHBG, CTX-I and CK-MB proteins.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65
* Proximal femur fracture (Group 1)

Exclusion Criteria:

* neoplasmatic history in the anamnesis,
* prevalent fracture
* mental illness
* immune disease affecting protein balance

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients admitted to the Department of Orthopaedics and Rehabilitation (due to proximal femur fracture) or to the Department of Internal Medicine (due to exacerbation of chronic disease process). The citizens of Warsaw in age over 65 who meet inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Serum concentration of SHBG and comparison between intervention groups | (Group 1) At the day of the admission to the Department of Orthopaedics and Rehabilitation prior the surgical treatment or (Group 2) at the day of the admission to the Department of Internal Medicine
Serum concentration of CTX-I and comparison between intervention groups | (Group 1) At the day of the admission to the Department of Orthopaedics and Rehabilitation prior the surgical treatment or (Group 2) at the day of the admission to the Department of Internal Medicine
Serum concentration of CK-MB and comparison between intervention groups | (Group 1) At the day of the admission to the Department of Orthopaedics and Rehabilitation prior the surgical treatment or (Group 2) at the day of the admission to the Department of Internal Medicine

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Othopedics and Rehabilitation, Medical University of Warsaw, Warsaw, Poland